CLINICAL TRIAL: NCT00004107
Title: Phase I/II Radioimmunotherapy of Non-Hodgkin's Lymphoma With High-Dose 90Y-Labeled Humanized LL2 Anti-CD-22 Antibody and Peripheral Blood Stem Cell Rescue
Brief Title: Radiolabeled Monoclonal Antibody Therapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Lymphoma or Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert M Sharkey, GSCC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067327; R01CA067026 (NIH); CMMI-C-037B-97; UPCC-1499; NCI-H99-0040
Record Dates: First submitted 1999-12-10; First posted 2004-04-16 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenstrom macroglobulinemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; B-cell adult acute lymphoblastic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation; Indium

INTERVENTIONS:
Biological: filgrastim — as prescribed by physician
Procedure: autologous bone marrow transplantation — 1-2 weeks before treatment
Procedure: peripheral blood stem cell transplantation — 1-2 weeks before treatment
Radiation: indium In 111 monoclonal antibody MN-14 — intravenous infusion over 30 min; single dose
Radiation: yttrium Y 90 epratuzumab — intravenous infusion over 30 min; single dose

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate cancer cells and deliver cancer-killing substances to them without harming normal cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by monoclonal antibody therapy used to kill cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody therapy plus peripheral stem cell transplantation in treating patients who have lymphoma or Waldenstrom's macroglobulinemia that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicity of radioimmunotherapy using high dose yttrium Y 90 humanized anti-CD22 monoclonal antibody LL2 (Y90 MOAB hLL2) followed by autologous peripheral blood stem cell transplantation in patients with B cell lymphomas or Waldenstrom's macroglobulinemia. II. Determine the organ and tumor dosimetry for comparison to clinical measurement of toxicity and antitumor responses in these patients. III. Determine magnitude and duration of human anti-humanized LL2 antibody (HAhLL2) or anti-DOTA response in these patients. IV. Evaluate the extent and duration of antitumor response to this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients are stratified according to prior treatment (high dose chemotherapy with transplantation vs low dose chemotherapy with radioimmunotherapy (RAIT) vs low dose chemotherapy without RAIT). Patients receive filgrastim (G-CSF) subcutaneously (SC) daily for 5 days and undergo harvest of peripheral blood stem cells (PBSC). If an adequate number of CD34+ cells are not harvested, autologous bone marrow may be used. Patients undergo pretherapy imaging with indium In 111 monoclonal antibody MN-14 (In111-MN-14) IV on day -7. If at least 1 tumor site is targeted, patients receive high dose yttrium Y 90 humanized anti-CD22 monoclonal antibody LL2 (Y90 MOAB hLL2) IV for up to 50 minutes on day 0. PBSC or bone marrow is reinfused approximately 7-14 days following infusion of Y90 MOAB hLL2. Patients also receive G-CSF SC daily until 3 days after blood counts have recovered. Cohorts of 3-6 patients receive escalating doses of Y90 MOAB hLL2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed weekly for 2 months, monthly for 6 months, and then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 12-24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven B cell lymphoma of one of the following types: Any histologic grade of non-Hodgkin's lymphoma Chronic lymphocytic leukemia CD22 positive acute lymphocytic leukemia Waldenstrom's macroglobulinemia Must have failed at least 1 standard therapy Autologous peripheral blood stem cells (PBSC) or bone marrow available Bone marrow involvement allowed if: Autologous bone marrow or PBSC with no greater than 5% tumor involvement available Radiation dose to marrow no greater than 3,000 cGy until 6 patients have been safely treated at that dose level At least 1 confirmed site of tumor targeted by pretherapy indium In 111 monoclonal antibody MN-14 imaging No brain metastases

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: Karnofsky 70-100% ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL AST and alkaline phosphatase less than 1.5 times upper limit of normal (ULN) in the absence of bone involvement Renal: Creatinine less than 1.5 times ULN Cardiovascular: Ejection fraction at least 50% Pulmonary: DLCO at least 60% of predicted Forced vital capacity at least 60% of predicted Other: No severe anorexia, nausea, or vomiting No concurrent significant medical complications that would preclude study participation Not pregnant Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior radioimmunotherapy AND high dose chemotherapy Chemotherapy: No prior high dose chemotherapy AND radioimmunotherapy At least 4 weeks since other prior chemotherapy and recovered Endocrine therapy: At least 2 weeks since prior corticosteroids and recovered Radiotherapy: No prior radioimmunotherapy AND high dose chemotherapy At least 4 weeks since prior radiotherapy to index lesion No prior radiotherapy to greater than 25% of any critical organ (e.g., lung, liver, kidneys) No prior total body irradiation Surgery: At least 4 weeks since prior major surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1998-02; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (4):
- United States (4):
  - Garden State Cancer Center, Belleville, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania